CLINICAL TRIAL: NCT02148900
Title: Development of a Blood Test for Marfan Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shriners Hospitals for Children (Other)
Collaborators: Oregon Health and Science University (Other); University of Utah (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lynn Y. Sakai, Ph.D., Sr. Investigator, Shriners Hospitals for Children
Other Study IDs: 79135
Record Dates: First submitted 2014-05-23; First posted 2014-05-28 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Marfan Syndrome; Marfan Related Disorders; Control Subjects
Keywords: Marfan syndrome; blood test; aortic root size; Marfan related disorders
MeSH Terms: conditions — Marfan Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma Frozen Cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Marfan: Diagnosis of Marfan syndrome, according to Ghent criteria.
- Marfan Related Disorders: Diagnosis of Loeys-Dietz syndrome, vascular Ehlers-Danlos syndrome, or Familial Thoracic Aortic Aneurysm and Dissection.
- Control Subjects: Unaffected by Marfan or Marfan related disorders.

SUMMARY:
The objective of this study is to determine whether a simple blood test can be a useful clinical tool for monitoring aortic disease in Marfan syndrome and Marfan-related disorders.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether increased quantitites of circulating microfibril fragments, measured with a simple blood test, are associated with aortic root size and increased growth of the aortic root in Marfan syndrome and related disorders. The secondary objectives of this study are to: (1) Determine a Marfan "signature" profile of circulating microfibril fragments. (2) Determine if high concentrations of fibrillin-1 fragments are associated with large aortic root diameters. (3) Determine which fibrillin-1 fragments are good biomarkers for aortic root growth and size in Marfan syndrome. (4) Determine the relation between fibrillin-1, aortic root diameter, and medical and lifestyle factors reported on questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-26 years of age for all participants
* Diagnosis of Marfan syndrome, Loeys-Dietz syndrome, vascular Ehlers-Danlos syndrome, or Familial Thoracic Aortic Aneurysm and Dissection for inclusion in Marfan and Marfan-related disorders groups
* Diagnosis of unaffected by Marfan syndrome and Marfan-related disorders for inclusion in control group
* Able and willing to sign informed consent/assent
* Signed HIPPA compliant research authorization

Exclusion Criteria:

* Other known cardiovascular disorder for unaffected controls

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population includes 3 groups: (1) individuals with Marfan syndrome; (2) individuals with Marfan-related disorders; (3) unaffected controls. Both genders, ages 4 to 26, will be included. Geographic locations will include the Pacific Northwest, Texas, and the Salt Lake City/Denver areas.
Sampling Method: Probability Sample
Enrollment: 336 (Estimated)
Dates: Start 2013-05; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
microfibril fragments | measured yearly over 5 years
  Plasma will be tested using sandwich ELISAs and standard curves to quantitate fragments of fibrillin-1, fibrillin-2, and fibulin-4.

SECONDARY OUTCOMES:
Aortic root growth | yearly for five years
  Aortic root growth will be correlated with concentrations of circulating microfibril fragments.

OTHER OUTCOMES:
medical and lifestyle issues | yearly for five years
  Information from questionnaires will be associated with aortic root growth and concentrations of circulating microfibril fragments.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Y. Sakai, Ph.D., Principal Investigator — Shriners Hospitals for Children
Locations (5):
- United States (5):
  - Lurie Childrens Hospital, Chicago, Illinois
  - University of Nebraska, Omaha, Nebraska
  - Oregon Health & Science University, Portland, Oregon
  - Shriners Hospital for Children, Portland, Oregon
  - University of Texas at Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No